CLINICAL TRIAL: NCT06416852
Title: A Multicenter, Open, Non-inferiority Phase III Clinical Study to Evaluate the Efficacy of 18F-Alfatide Injection PET/CT Compared With 18F-FDG PET/CT in the Diagnosis of Lymph Node Metastasis in Non-small Cell Lung Cancer
Brief Title: Clinical Study of 18F-Alfatide Injection PET/CT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yantai LNC Biotechnology Singapore PTE. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-Alfatide-003
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer NSCLC
MeSH Terms: interventions — alfatide II; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Alfatide and 18F-FDG Injection (Experimental): The study is designed as a self-controlled trial, in which participants will be injected and scanned with two drugs.
  Interventions: Drug: 18F-Alfatide Injection; Drug: 18F-FDG Injection

INTERVENTIONS:
Drug: 18F-Alfatide Injection — A single dose of (0.1~0.15）±0.015 mCi/kg IV injection of 18F-Alfatide. The patients will be intravenously injected with 18F-Alfatide Injection and undergo PET/CT scan at 60 min±10 min after the injection.
Drug: 18F-FDG Injection — A single dose of 5～10mCi IV injection of 18F-FDG. The patients will be intravenously injected with 18F-FDG Injection and undergo PET/CT scan at 40 min±10 min after the injection.

SUMMARY:
This is a multicenter, open, non-inferiority Phase III clinical study to evaluate the efficacy of 18F-Alfatide Injection PET/CT compared with 18F-FDG PET/CT in the diagnosis of lymph node metastasis in non-small cell lung cancer.

This trial will include 428 patients with non-small cell lung cancer confirmed by imaging, histopathology and/or cytology or highly suspected by investigators, suspected lymph node metastasis and proposed radical surgery and lymph node dissection. Eligible subjects will receive 18F-Alfatide Injection PET/CT and 18F-FDG PET/CT scans within 1 week. Subjects will undergo relevant security checks before and after each scan. The subjects underwent radical surgery and lymph node dissection within 2 weeks of completing both scans, and the obtained lymph nodes were pathologically examined as the gold standard to compare the diagnostic efficacy of 18F-Alfatide versus 18F-FDG for lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects understand the clinical trial procedure and sign the informed consent in person;
2. Patients with non-small cell lung cancer confirmed or highly suspected by investigators based on prior history, imaging, histopathology, and/or cytology, suspected lymph node metastasis and proposed radical surgery and lymph node dissection;
3. Over 18 years old (including 18 years old);
4. ECOG function status score 0~1 points ;
5. Expected survival > 3 months.

Exclusion Criteria:

1. Known allergic history to 18F-Alfatide Injection and 18F-FDG injection or its excipients;
2. Patients who cannot tolerate intravenous drug administration (such as needle fainting and blood fainting history);
3. Patients who are not suitable for PET or cannot complete PET or other imaging tests due to special reasons, including claustrophobia and radiophobia;
4. Workers who need to be exposed to radioactive conditions for a long time;
5. Patients with renal insufficiency were defined as the standard endogenous creatinine clearance (Ccr) estimated by the Cockcroft-Gault formula <60 ml/min, Ccr(ml/min)=[(140-age)× body weight (kg)]/[72×Scr(mg/dl)], and the calculated result for females was 0.85;
6. Fasting blood glucose level more than 7.0 mmol/L;
7. There are serious infections that cannot be controlled before screening;
8. Any serious disease that cannot be controlled, such as severe heart dysfunction (such as unstable angina pectoris, myocardial infarction, heart failure, etc.), a large number of pleural effusion patients, patients with mental illness, etc.;
9. Previously diagnosed with other malignant tumors, except in the following cases:

   * Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing prior to enrollment in the study);
   * Carcinoma in situ of cervical or breast cancer with curative treatment and no signs of recurrence for at least 3 years prior to the study;
   * The primary malignancy has been completely removed and in complete remission for ≥5 years.
10. Participants who had participated in clinical trials of radiopharmaceuticals within 1 year before screening;
11. Participating in other interventional clinical trials within 1 month before screening;
12. Poor general condition, heart, lung, liver, kidney, brain and other vital organs can not tolerate surgery;
13. Those who had a birth plan during the trial and within 1 year after the completion of the trial, or the subjects and their spouses did not agree to take strict contraceptive measures during the trial and within 6 months after the completion of the trial (using condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.);
14. Pregnant or lactating female subjects;
15. Subjects with poor compliance or other factors deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity evaluation of 18F-Alfatide Injection PET/CT compared with 18F-FDG PET/CT | Through study completion, assessed up to 2 years
  To evaluate the sensitivity and specificity of 18F-Alfatide Injection PET/CT in the diagnosis of lymph node metastasis in non-small cell lung cancer compared with 18F-FDG PET/CT.All subjects in this study underwent 18F-Alfatide PET-CT and 18F-FDG PET-CT examination within one week, radical surgery and lymph node dissection within two weeks after the completion of the two scanning images, and pathological examination of the obtained lymph nodes was used as the gold standard.

SECONDARY OUTCOMES:
Accuracy, positive predictive value and negative predictive value evaluation of 18F-Alfatide Injection PET/CT compared with 18F-FDG PET/CT | Through study completion, assessed up to 2 years
  To evaluate the accuracy, positive predictive value and negative predictive value of 18F-Alfatide Injection PET/CT in the diagnosis of lymph node metastasis in non-small cell lung cancer compared with 18F-FDG PET/CT.All subjects in this study underwent 18F-Alfatide PET-CT and 18F-FDG PET-CT examination within one week, radical surgery and lymph node dissection within two weeks after the completion of the two scanning images, and pathological examination of the obtained lymph nodes was used as the gold standard
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, assessed up to 2 years
  To evaluate the safety of 18F-Alfatide Injection PET/CT in the diagnosis of lymph node metastasis in non-small cell lung cancer compared with 18F-FDG PET/CT.The safety will be assessed by the number and percentage of patients with adverse events; Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No